CLINICAL TRIAL: NCT00203736
Title: Open Label Drug Study (With Single and Parallel Group Components) to Evaluate Combination Antimalarial Therapy for Efficacy, Gametocyte Carriage and Molecular Markers Associated With SP Resistance in Uncomplicated Plasmodium Falciparum Infections
Brief Title: A Randomised Efficacy Study of Combination Antimalarials to Treat Uncomplicated Malaria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: World Health Organization (Other); Medical Research Council, South Africa (Other); Global Fund (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SEACAT 01 Am 4 (RCT)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2006-11-16 (Estimated); Status verified 2005-08

CONDITIONS: Malaria
Keywords: Malaria; Efficacy; Pharmacokinetic; Gametocyte; Molecular Markers; Sulfadoxine-pyrimethamine; Artesunate; Artemisinin
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination; Artesunate

INTERVENTIONS:
Drug: Sulfadoxine-pyrimethamine
Drug: Artesunate plus sulfadoxine-pyrimethamine

SUMMARY:
The purpose of this study is to compare the efficacy of sulfadoxine-pyrimethamine plus artesunate with that of sulfadoxine-pyrimethamine on its own for the treatment of uncomplicated malaria.

DETAILED DESCRIPTION:
Resistance of Plasmodium falciparum to anti-malarial drugs is a serious impediment to malaria control. In the South East African Combination Anti-malarial Therapy (SEACAT) evaluation, there is an evaluation of the phased introduction of combination anti-malarial therapy (CAT) in Mozambique, Swaziland and South Africa. In order to facilitate formulation of effective regional drug policy and provide a database for decision-making on the implementation of CAT, it is essential that the in vivo response to CAT be investigated. This will be achieved through the SEACAT 01 protocol which is a component of the SEACAT evaluation described in another file on this website. However, in selected Mozambique sites where the intensity of malaria transmission is high, a direct parallel group comparison of monotherapy (SP) with CAT (artesunate, AS, plus SP) will be conducted according to a specific amendment (Amendment 4) to the SEACAT 01 protocol. Amendment 4 is presented in this separate file on the website for clarity.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, older than 12 months.
* Weight > 10 kg.
* Diagnoses of uncomplicated acute P. falciparum malaria parasitaemia of up to 500 000 asexual parasite/mcl blood with axillary temperature of greater than and equal to 37.50C or history of fever.
* Documented informed consent.
* Lives close enough to the health centre for reliable follow up.

Exclusion Criteria:

* Has received anti-malarial treatment in the past 7 days.
* Is infected with other malarial species (such subjects will be excluded retrospectively).
* Severely ill (based on WHO Criteria for severe malaria ) or if patient is considered, in the opinion of the investigator or designee, to have moderately severe malaria (e.g. prostrate, repeated vomiting, dehydrated).
* Has received cotrimoxazole or chloramphenicol in the past 7 days.
* History of G6PD deficiency.
* Is pregnant.
* Has a history of allergy to any sulphonamide (for SP) or artemisinin derivative (for artesunate and co-artemether).

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240
Dates: Start 2003-01; Study Completion 2003-10

PRIMARY OUTCOMES:
Therapeutic efficacy defined as: Adequate Clinical and Parasitological Response (ACPR), Early Treatment Failure (ETF), Late Treatment Failure (LTF), defined as Late Clinical Failure (LCF) and Late Parasitological Failure (LPF)
Sensitive or parasitological failure (RI, early and late, RII, RIII)
Parasitological failures will be classified as recrudescence or re-infection (or indeterminate) using GLURP and MSP I & II markers
Parasite clearance time
Fever clearance time

SECONDARY OUTCOMES:
Association between study treatment and gametocyte carriage
Pharmacokinetics by measurement of whole blood levels of Sulfadoxine and Pyrimethamine
Correlation of frequency of DHFR and DHPS mutations with parasitological outcome
Tolerability by describing adverse events and changes in haematological parameters
Capacity by describing the training and development of study teams

CONTACTS AND LOCATIONS:
Overall Officials: Karen Barnes, MBChB, Principal Investigator — University of Cape Town
Locations (2):
- Mozambique (2):
  - Catuane Clinic, Catuane, Matutuine
  - Namaacha Clinic, Namaacha, Namaacha

REFERENCES:
- [Derived] Allen EN, Little F, Camba T, Cassam Y, Raman J, Boulle A, Barnes KI. Efficacy of sulphadoxine-pyrimethamine with or without artesunate for the treatment of uncomplicated Plasmodium falciparum malaria in southern Mozambique: a randomized controlled trial. Malar J. 2009 Jun 26;8:141. doi: 10.1186/1475-2875-8-141. PMID 19558654